CLINICAL TRIAL: NCT05286554
Title: Impact of Addition of Gonadotropin Releasing Hormone Agonist to Luteal Phase Support on Antagonist ICSI Cycles
Brief Title: Addition of Gonadotropin Releasing Hormone Agonist to Luteal Phase Support
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201599
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2022-03

CONDITIONS: Female Infertility
Keywords: luteal phase support, ICSI, gonadotropin releasing hormone agonist
MeSH Terms: conditions — Infertility, Female | interventions — Gonadotropin-Releasing Hormone; Triptorelin Pamoate; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Will receive routine LPS and additional single GnRH-a bolus, triptorelin 0.1 mg subcutaneous injection on the 6th day after oocyte retrieval.
  Interventions: Drug: gonadotropin releasing hormone-agonist; Drug: Progesterone
- Group 2 (Experimental): Will receive routine LPS and additional multiple mid-luteal GnRH-a, triptorelin 0.1 mg subcutaneous injection on the 5th, 7th and 9th days after oocyte retrieval.
  Interventions: Drug: gonadotropin releasing hormone-agonist; Drug: Progesterone
- Group 3 (Control) (Active Comparator): Will receive the routine LPS without GnRH-a
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: gonadotropin releasing hormone-agonist — subcutaneous injection
  Other Names: triptorelin 0.1 mg
  Arms: Group 1; Group 2
Drug: Progesterone — vaginal suppositories (400 mg twice daily) starting on the day after oocyte retrieval and will be continued till pregnancy assessed by serum β-HCG 15 days after ICSI, and if pregnant, for 10 weeks of gestation.
  Other Names: cyclogest

SUMMARY:
Hormonal milieu during implantation is crucial to embryo-endometrium interaction and to the viability of the conceptus. Alterations in the peri-implantation environment are considered to impair perinatal outcomes in intracytoplasmic sperm injection (ICSI) therapy. GnRH-a is a new and promising modality for LPS. Regimens for using GnRH-a in LPS, including single mid-luteal bolus or the addition of a GnRH-a to progesterone supplementation, have been recently suggested. The aim of this study is to evaluate the impact of addition of mid-luteal single-dose or multiple-dose GnRH agonist to the routine luteal phase support in patients undergoing ICSI cycles using GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≤ 38 years.
2. BMI ≤ 30.
3. Basal follicle stimulating hormone (FSH) level ≤ 10 IU/L.
4. Anti-Müllerian hormone (AMH): ≤ 5 ng/ml.

Exclusion Criteria:

1. Endometriosis.
2. Polycystic ovarian syndrome (PCOS).
3. Uterine pathology or anomaly.
4. Evidence of hydrosalpinx by hysterosalpingography or ultrasound.
5. Comorbidities: Diabetes mellitus, hypertension, immune diseases.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 2 weeks after positive pregnancy test
  Calculated as the number of clinical pregnancies (Presence of an intrauterine gestational sac with embryonic cardiac activity observed by vaginal ultrasound) divided by the number of embryo transfer procedures.

SECONDARY OUTCOMES:
Implantation rate | 2 weeks after positive pregnancy test
  the ratio of the number of gestational sacs detected by sonography to the total number of embryos transferred.
Multiple pregnancy rate | 8 weeks of gestation
  The percentage of pregnancies with more than one fetus
Serum β-human chorionic gonadotropin (β-HCG) concentration | 15 days after ICSI
  In milli-International unit/ml on day 15 after ICSI

CONTACTS AND LOCATIONS:
Overall Officials: Mervat Sheikh El-arab, PhD, Principal Investigator — Alexandria Univsersity; Ahmed Abdel Aziz, PhD, Study Director — Alexandria Univsersity
Locations (1):
- Alexandria University, Alexandria, Alexandria Governorate, Egypt

REFERENCES:
- [Background] de Ziegler D, Pirtea P, Andersen CY, Ayoubi JM. Role of gonadotropin-releasing hormone agonists, human chorionic gonadotropin (hCG), progesterone, and estrogen in luteal phase support after hCG triggering, and when in pregnancy hormonal support can be stopped. Fertil Steril. 2018 May;109(5):749-755. doi: 10.1016/j.fertnstert.2018.03.006. PMID 29778367
- [Background] Thomsen LH, Kesmodel US, Andersen CY, Humaidan P. Daytime Variation in Serum Progesterone During the Mid-Luteal Phase in Women Undergoing In Vitro Fertilization Treatment. Front Endocrinol (Lausanne). 2018 Mar 19;9:92. doi: 10.3389/fendo.2018.00092. eCollection 2018. PMID 29615975
- [Background] Shoham G, Leong M, Weissman A. A 10-year follow-up on the practice of luteal phase support using worldwide web-based surveys. Reprod Biol Endocrinol. 2021 Jan 26;19(1):15. doi: 10.1186/s12958-021-00696-2. PMID 33499875
- [Background] Wang NF, Bungum L, Skouby SO. What is the optimal luteal support in assisted reproductive technology? Horm Mol Biol Clin Investig. 2021 Feb 22;43(2):225-233. doi: 10.1515/hmbci-2020-0081. PMID 33609426
- [Background] Balasch J, Martinez F, Jove I, Cabre L, Coroleu B, Barri PN, Vanrell JA. Inadvertent gonadotrophin-releasing hormone agonist (GnRHa) administration in the luteal phase may improve fecundity in in-vitro fertilization patients. Hum Reprod. 1993 Jul;8(7):1148-51. doi: 10.1093/oxfordjournals.humrep.a138210. PMID 8408503
- [Background] Tesarik J, Hazout A, Mendoza C. Enhancement of embryo developmental potential by a single administration of GnRH agonist at the time of implantation. Hum Reprod. 2004 May;19(5):1176-80. doi: 10.1093/humrep/deh235. Epub 2004 Apr 7. PMID 15070873
- [Background] Tesarik J, Hazout A, Mendoza-Tesarik R, Mendoza N, Mendoza C. Beneficial effect of luteal-phase GnRH agonist administration on embryo implantation after ICSI in both GnRH agonist- and antagonist-treated ovarian stimulation cycles. Hum Reprod. 2006 Oct;21(10):2572-9. doi: 10.1093/humrep/del173. Epub 2006 Aug 22. PMID 16926261
- [Background] Fusi FM, Arnoldi M, Bosisio C, Lombardo G, Ferrario M, Zanga L, Galimberti A, Capitanio E. Ovulation induction and luteal support with GnRH agonist in patients at high risk for hyperstimulation syndrome. Gynecol Endocrinol. 2015;31(9):693-7. doi: 10.3109/09513590.2015.1025379. Epub 2015 Aug 31. PMID 26527503
- [Background] Ma X, Du W, Hu J, Yang Y, Zhang X. Effect of Gonadotrophin-Releasing Hormone Agonist Addition for Luteal Support on Pregnancy Outcome in vitro Fertilization/Intracytoplasmic Sperm Injection Cycles: A Meta-Analysis Based on Randomized Controlled Trials. Gynecol Obstet Invest. 2020;85(1):13-25. doi: 10.1159/000501204. Epub 2019 Aug 16. PMID 31422404
- [Background] Aboulghar MA, Marie H, Amin YM, Aboulghar MM, Nasr A, Serour GI, Mansour RT. GnRH agonist plus vaginal progesterone for luteal phase support in ICSI cycles: a randomized study. Reprod Biomed Online. 2015 Jan;30(1):52-6. doi: 10.1016/j.rbmo.2014.09.017. Epub 2014 Oct 13. PMID 25456166
- [Background] Isikoglu M, Ozgur K, Oehninger S. Extension of GnRH agonist through the luteal phase to improve the outcome of intracytoplasmic sperm injection. J Reprod Med. 2007 Jul;52(7):639-44. PMID 17847764
- [Background] Martins WP, Ferriani RA, Navarro PA, Nastri CO. GnRH agonist during luteal phase in women undergoing assisted reproductive techniques: systematic review and meta-analysis of randomized controlled trials. Ultrasound Obstet Gynecol. 2016 Feb;47(2):144-51. doi: 10.1002/uog.14874. Epub 2015 Dec 30. PMID 25854891
- [Background] Qu D, Li Y. Multiple-dose versus single-dose gonadotropin-releasing hormone agonist after first in vitro fertilization failure associated with luteal phase deficiency: A randomized controlled trial. J Int Med Res. 2020 Jun;48(6):300060520926026. doi: 10.1177/0300060520926026. PMID 32495663